CLINICAL TRIAL: NCT04143737
Title: Community-Based Lifestyle Intervention for Primary and Secondary Prevention of Diabetes in Arab Women in East-Jerusalem, A Quasi-experimental Study.
Brief Title: Community-Based Lifestyle Intervention for Primary and Secondary Prevention of Diabetes in Arab Women in East-Jerusalem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZU456-HMO-CTIL
Record Dates: First submitted 2018-11-29; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2017-06

CONDITIONS: Diabetes; Cardiovascular Diseases; Health Behavior
Keywords: Community-based intervention; Arab women; East jerusalem; Diabetes prevention; Lifestyle intervention; Quasi-Experiment
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): 38 women participated in the intervention group which was located in a community center in Zur-Baher neighborhood. The intervention consisted of 20 weekly sessions on nutrition, physical activity, stress management skills, and self-monitoring. All taught by professional facilitators (nutritionists, exercise trainers, health coaches, and psychotherapists). Baseline data was collected
  Interventions: Behavioral: Healthy lifestyle intervention
- Control (No Intervention): 22 women participated in the control group. They were recruited from a community center in the old city of Jerusalem and did not receive any intervention. Baseline data was collected.

INTERVENTIONS:
Behavioral: Healthy lifestyle intervention — 38 women participated in the intervention group which was located in a community center in Zur-Baher neighborhood. The intervention consisted of 20 weekly sessions on nutrition, physical activity, stress management skills, and self-monitoring. All taught by professional facilitators (nutritionists, exercise trainers, health coaches, and psychotherapists). Baseline data was collected
  Arms: Intervention

SUMMARY:
Given the extremely high incidence of diabetes in Arab women and the current lack of interventions, all non-diabetic women can be considered "at risk" and warrant secondary prevention. Creating an effective community-based primary and secondary diabetes prevention program has the potential for nationwide reduction of health disparities for Arab women.

The purpose of this study was to investigate the effectiveness of a lifestyle intervention in reducing risky health behaviors and thus reducing modifiable risk factors associated with diabetes and cardiovascular diseases, through dietary modification, adherence to healthy low-caloric, low-fat diet and engaging in physical activity.

DETAILED DESCRIPTION:
Given the extremely high incidence of diabetes in Arab women and the current lack of interventions, all non-diabetic women can be considered "at risk" and warrant secondary prevention.

The purpose of this study was to investigate the effectiveness of lifestyle intervention in reducing risky health behaviors and thus reducing modifiable risk factors associated with diabetes and cardiovascular diseases, through dietary modification, adherence to healthy low-caloric, low-fat diet and engaging in physical activity.

Methods: The invistigators will conduct a quasi-experimental, pre-post intervention study between to investigate the effectiveness of community based intervention to change lifestyle habits and consequently reduce the modifiable risk factors for developing diabetes at all levels of prevention. All members of two targeted Arab women's community centers in East-Jerusalem will be invited to participate in the study. Potential participants will be interviewed for eligibility (over age 25, able to commit to the intervention timetable, and precluding pregnancy or serious mental and physical illness).

Participants who will be included in the control group will not receive any intervention. The intervention group will be located in one community center in Zur-Baher neighborhood, and the control group will be located in one community center in the old city of Jerusalem.

Data will be collected from both groups. Intervention: The Community-Based Lifestyle Intervention (CBLI) was developed based on the gold standard Diabetes Prevention Program (DPP) and adapting all intervention components to the specific culture, language, gender, and religious sensitivities of Palestinian female society. The intervention consisted of 20 weekly sessions and will be taught by professional facilitators (nutritionists, exercise trainers, health coaches, and psychotherapists). The DPP's lifestyle curriculum includes sessions on nutrition, physical activity, stress management skills, and self-monitoring and was culturally adapted, translated into Arabic, and gender tailored.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 and above
* Able to commit to the program timetable

Exclusion Criteria:

* Age younger than25
* Unable to commit to the intervention timetable
* Pregnant with expected delivery during the intervention
* Women with serious mental or physical illness

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Adherence to Mediterranean diet | 6 months after intervention initiation
  Adherence to Mediterranean Diet- Eating behaviors will be assessed through self-reported questionnaire adapted from the Attica study. The questions include an assessment of daily average consumption of whole grains, vegetables, fruits, legumes, and low-fat dairy products. The questionnaire includes also food items assessing the consumption of western diet including sweets, sweet drinks and salty snacks. These questions were adapted from the following study: "A Western dietary pattern is associated with higher blood pressure in Iranian adolescents." European Journal of Nutrition 2017 Feb:56(1)399-408.
Change in average daily steps- measured by Pedometer | 6 months after intervention initiation
  The participants in the intervention group were given a pedometer and weekly step data were collected by the research team.

SECONDARY OUTCOMES:
Change in body Mass Index (BMI) | 6 months after intervention initiation
  BMI will be calculated by measuring weight and height for each participant. weight will be measured in kilograms. Height was measured to the nearest 0.1 cm. Body Mass Index (BMI) will be calculated using the formula of weight in kg divided by height in m2 (kg/m2).
Change in Plasma levels of Hemoglobin A1c (HbA1c) | 6 months after intervention initiation
  measured using capillary whole blood obtained on finger stick, through a cartridge-based latex agglutination inhibition assay through finger stick on the Cobas B101 point of care device
Change in Plasma levels of Glucose, HDL, LDL, triglycerides, and total cholesterol | 6 months after intervention initiation
  The participants will be referred to their national health insurance in order to conduct a blood test for plasma levels of HDL, LDL, triglycerides, and total cholesterol
Change in Blood pressure (BP) | 6 months after intervention initiation
  Will be measured using standard procedures with an electronic BP apparatus and the recorded measurement is the average of 2 measurements taken in the seated position
Change in Cardiovascular disease knowledge | 6 months after intervention initiation
  Will be assessed through self report questionnaire based on the American Heart Association's knowledge survey items
Change in Leadership self-efficacy scale | 6 months after intervention initiation
  Leadership self-efficacy will be assessed through self report questionnaire. This questionnaire was adapted from a scale used in previous study by the Brookdale Institute in Israel, with similar objectives of empowering and promoting female lay health leaders in the community to advance women's health. The questionnaire consists of 9 items. Participants were asked to rate their level of confidence that they can perform the tasks defined by the leadership component objectives. Respondents select from a 4-point scale varying from 1 = a little confident to 4 = very confident. The sub-scales will be summed and average score will be calculated. higher values represent a better outcome.

IPD SHARING:
Plan to Share IPD: Yes
Plan is to share de-identified IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be available with publication
Access Criteria: GCP certification and review of appropriate research interest

REFERENCES:
- [Background] Ackermann RT. Bridging the why and the how of clinical-community integration. Am J Prev Med. 2013 Oct;45(4):526-9. doi: 10.1016/j.amepre.2013.07.003. No abstract available. PMID 24050431
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Chiuve SE, Cook NR, Shay CM, Rexrode KM, Albert CM, Manson JE, Willett WC, Rimm EB. Lifestyle-based prediction model for the prevention of CVD: the Healthy Heart Score. J Am Heart Assoc. 2014 Nov 14;3(6):e000954. doi: 10.1161/JAHA.114.000954. PMID 25398889
- [Background] Chan JC, Malik V, Jia W, Kadowaki T, Yajnik CS, Yoon KH, Hu FB. Diabetes in Asia: epidemiology, risk factors, and pathophysiology. JAMA. 2009 May 27;301(20):2129-40. doi: 10.1001/jama.2009.726. PMID 19470990
- [Background] Fianu A, Bourse L, Naty N, Le Moullec N, Lepage B, Lang T, Favier F. Long-Term Effectiveness of a Lifestyle Intervention for the Primary Prevention of Type 2 Diabetes in a Low Socio-Economic Community--An Intervention Follow-Up Study on Reunion Island. PLoS One. 2016 Jan 5;11(1):e0146095. doi: 10.1371/journal.pone.0146095. eCollection 2016. PMID 26731676
- [Background] Kalter-Leibovici O, Chetrit A, Lubin F, Atamna A, Alpert G, Ziv A, Abu-Saad K, Murad H, Eilat-Adar S, Goldbourt U. Adult-onset diabetes among Arabs and Jews in Israel: a population-based study. Diabet Med. 2012 Jun;29(6):748-54. doi: 10.1111/j.1464-5491.2011.03516.x. PMID 22050554
- [Background] Idilbi NM, Barhana M, Milman U, Carel RS. [Diabetes mellitus and cancer: the different expression of these diseases in Israeli Arabs and Jews]. Harefuah. 2012 Nov;151(11):625-8, 654. Hebrew. PMID 23367733
- [Background] Panagiotakos DB, Chrysohoou C, Pitsavos C, Stefanadis C. Association between the prevalence of obesity and adherence to the Mediterranean diet: the ATTICA study. Nutrition. 2006 May;22(5):449-56. doi: 10.1016/j.nut.2005.11.004. Epub 2006 Feb 2. PMID 16457990
- [Background] Hojhabrimanesh A, Akhlaghi M, Rahmani E, Amanat S, Atefi M, Najafi M, Hashemzadeh M, Salehi S, Faghih S. A Western dietary pattern is associated with higher blood pressure in Iranian adolescents. Eur J Nutr. 2017 Feb;56(1):399-408. doi: 10.1007/s00394-015-1090-z. Epub 2015 Nov 3. PMID 26534856